CLINICAL TRIAL: NCT02602652
Title: Immunogenicity of a Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) as a Booster Dose After a Primary Vaccination With SA14-14-2 Vaccine in Thai Children
Brief Title: Immunogenicity of a JE-CV as a Booster Dose After a Primary Vaccination With SA14-14-2 Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB456/56
Record Dates: First submitted 2015-10-12; First posted 2015-11-11 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Japanese Encephalitis
Keywords: geometric mean titer; seroprotection; live attenuated chimeric JE vaccine; JE-CV; SA14-14-2 vaccine
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- a live attenuated chimeric JE vaccine (Experimental): Children were received JE-CV as a booster dose after vaccinated with SA14-14-2 vaccine as a first dose regimen 12-24 months before.
  Interventions: Biological: a live attenuated chimeric JE vaccine

INTERVENTIONS:
Biological: a live attenuated chimeric JE vaccine — The study included 2 visits (D0 and D28). At the first visit (D0), children were enrolled, collected the blood sample for evaluate the baseline immune status and given a JE-CV as a booster dose. After vaccination, children were observed for 30 minutes to monitor any immediate adverse events. Parents were given a digital thermometer for axillary temperature measurement, a ruler for measuring injection site reactions and a diary card for recording a solicited injection site and systemic reactions.
  At the second visit (D28), blood samples were collected for evaluate the immunogenicity.
  Other Names: Japanese Encephalitis Chimeric Virus vaccine

SUMMARY:
The objective of this study is to measured the Geometric mean titer (GMT) of Japanese Encephalitis neutralizing antibody and proportion of seroprotection among the children who received a booster dose of JE-CV after the first dose of SA14-14-2 vaccine.

DETAILED DESCRIPTION:
Study design: This open label clinical trial in 50 children aged 1-5 years, was conducted at King Chulalongkorn Memorial Hospital in Thailand. The protocol was approved by the Institutional Review Board of Chulalongkorn University, and the study was performed in accordance with Declaration of Helsinki, International Conference on Harmonization Good Clinical Practice, the European Directive 2001/20/EC, and written informed consent was obtained from parents or a legally acceptable representative before enrolment.

Vaccines: JE-CV was manufactured by Sanofi Pasteur Biologics Co., USA., and reconstituted using 0.4% sodium chloride diluent for injection; each dose 0.5 ml contained 4.0-5.8 log10 plaque forming units of virus Serology: JE neutralizing antibody levels were assessed using a PRNT50 assay. The final end point neutralization titer is the inverse of the highest serial dilution of serum that can neutralize ≥ 50% of JE challenge virus. Testing was performed at Focus Diagnostics Inc. using JE-CV as a challenge virus.

Statistical methods: sample size was calculated based on historical data from JE15 study, at month 24 after first dose of JE-CV, the GMT of JE neutralizing antibody was 39.4 (95% CI 33.7 to 46.0) and increase to 2242 (95% CI 1913, 2628) at day 28 post JE-CV booster dose. On the assumption that children who received SA14-14-2 vaccine and subsequently get one booster dose of JE-CV at 12-24 months later will have GMT of at least 1040, with 80% power and alpha 0.05, data at least 43 children need to be collected. When accounted for 15% of children who might loss to follow-up or cannot get adequate blood sample, 50 children should be enrolled.

The per-protocol population will be used for the main immunogenicity analyses. For the main parameters, 95% confidence intervals (CIs) of point estimates will be calculated using the normal approximation for quantitative data and the exact binomial distribution for proportions. The point estimates and their 95% CI of the following will be presented for each group of the Geometric Mean (GM) of neutralizing antibody on D0 and D28 and the percentage of subjects with neutralizing antibody >=10 at D0 and D28

ELIGIBILITY:
Inclusion Criteria:

1 Children aged 1 to <5 years on the day of inclusion

2. History of received 1 dose of SA14-14-2 vaccine 12-24 months prior to enrollment

3. In good general health at the time of inclusion

4. Provision of informed consent by the parent(s) or legal guardian(s)

Exclusion Criteria:

1. Receipt of blood or blood products in the past 3 months.
2. Acute febrile illness on the day of vaccination.( BT > 38 C)

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changing in geometric mean titer of JE neutralizing antibody at day 0 pre-vaccination and day 28 post vaccination. | day 0 pre-vaccination and day 28 post vaccination

SECONDARY OUTCOMES:
Proportion of children who had seroprotection at day 0 pre-vaccination and day 28 post vaccination | day 0 pre-vaccination and day 28 post vaccination
  seroprotection defined as titer ≥10

OTHER OUTCOMES:
JE-CV related adverse reaction | 28 days
  Solicited injection site reactions:
  * redness (in proportion of children)
  * swelling (in proportion of children)
  * pain (in proportion of children)
  Systemic solicited reactions: (measure in proportion of children)
  Unsolicited adverse reactions (measure in proportion of children)

CONTACTS AND LOCATIONS:
Overall Officials: Pakpoom Janewongwirot, md, Principal Investigator — Chulalongkorn University

REFERENCES:
- [Background] Feroldi E, Pancharoen C, Kosalaraksa P, Watanaveeradej V, Phirangkul K, Capeding MR, Boaz M, Gailhardou S, Bouckenooghe A. Single-dose, live-attenuated Japanese encephalitis vaccine in children aged 12-18 months: randomized, controlled phase 3 immunogenicity and safety trial. Hum Vaccin Immunother. 2012 Jul;8(7):929-37. doi: 10.4161/hv.20071. Epub 2012 Jul 1. PMID 22777096
- [Background] Feroldi E, Capeding MR, Boaz M, Gailhardou S, Meric C, Bouckenooghe A. Memory immune response and safety of a booster dose of Japanese encephalitis chimeric virus vaccine (JE-CV) in JE-CV-primed children. Hum Vaccin Immunother. 2013 Apr;9(4):889-97. doi: 10.4161/hv.23087. Epub 2013 Feb 26. PMID 23442823
- [Background] Chokephaibulkit K, Sirivichayakul C, Thisyakorn U, Sabchareon A, Pancharoen C, Bouckenooghe A, Gailhardou S, Boaz M, Feroldi E. Safety and immunogenicity of a single administration of live-attenuated Japanese encephalitis vaccine in previously primed 2- to 5-year-olds and naive 12- to 24-month-olds: multicenter randomized controlled trial. Pediatr Infect Dis J. 2010 Dec;29(12):1111-7. doi: 10.1097/INF.0b013e3181f68e9c. PMID 20856164
- [Background] Nasveld PE, Ebringer A, Elmes N, Bennett S, Yoksan S, Aaskov J, McCarthy K, Kanesa-thasan N, Meric C, Reid M. Long term immunity to live attenuated Japanese encephalitis chimeric virus vaccine: randomized, double-blind, 5-year phase II study in healthy adults. Hum Vaccin. 2010 Dec;6(12):1038-46. doi: 10.4161/hv.6.12.13057. Epub 2010 Dec 1. PMID 21150279
- [Background] Chotpitayasunondh T, Sohn YM, Yoksan S, Min J, Ohrr H. Immunizing children aged 9 to 15 months with live attenuated SA14-14-2 Japanese encephalitis vaccine in Thailand. J Med Assoc Thai. 2011 Aug;94 Suppl 3:S195-203. PMID 22043776
- [Background] Campbell GL, Hills SL, Fischer M, Jacobson JA, Hoke CH, Hombach JM, Marfin AA, Solomon T, Tsai TF, Tsu VD, Ginsburg AS. Estimated global incidence of Japanese encephalitis: a systematic review. Bull World Health Organ. 2011 Oct 1;89(10):766-74, 774A-774E. doi: 10.2471/BLT.10.085233. Epub 2011 Aug 3. PMID 22084515
- [Background] Centers for Disease Control and Prevention (CDC). Japanese encephalitis surveillance and immunization--Asia and the Western Pacific, 2012. MMWR Morb Mortal Wkly Rep. 2013 Aug 23;62(33):658-62. PMID 23965828
- [Derived] Janewongwirot P, Puthanakit T, Anugulruengkitt S, Jantarabenjakul W, Phasomsap C, Chumket S, Yoksan S, Pancharoen C. Immunogenicity of a Japanese encephalitis chimeric virus vaccine as a booster dose after primary vaccination with SA14-14-2 vaccine in Thai children. Vaccine. 2016 Oct 17;34(44):5279-5283. doi: 10.1016/j.vaccine.2016.09.005. Epub 2016 Sep 12. PMID 27628323